# **Study Protocol**

Official Title: Evaluation of PEEK Versus Titanium Bar Attachments with Implant-Assisted Mandibular Complete Overdenture Fabricated by CAD/CAM Technology

NCT Number: Not yet assigned

Document Date: February 20, 2024

Study Type:

Interventional (Clinical Trial)

# Study Design:

- Allocation: Randomized

- Intervention Model: Parallel Assignment

- Masking: None (Open Label)- Primary Purpose: Treatment

## Study Population:

- Total Sample Size: 12 patients

- Age Range: 40-60 years

- Inclusion Criteria:
- Completely edentulous mandibular arch
- Adequate bone quantity and quality for implant placement
- Class I maxilla-mandibular relationship
- Sufficient inter-arch space (≥25 mm)
- Good oral hygiene
- Exclusion Criteria:
- Systemic diseases affecting tissue healing
- History of radiation therapy in head/neck region
- Neurological or psychological disorders affecting oral hygiene
- Parafunctional habits
- Heavy smoking, alcoholism, or drug abuse

#### Study Groups / Interventions:

- Group I (Control): CAD/CAM Titanium bar attachment mandibular overdenture (6 patients)
- Group II (Study): CAD/CAM PEEK bar attachment mandibular overdenture (6 patients)

#### **Outcome Measures:**

#### Primary Outcome:

- Retention force of mandibular overdenture measured in Newtons using a digital force meter at insertion, 6 months, and 1 year

## **Secondary Outcomes:**

- Marginal bone loss around implants measured via digital periapical X-rays at insertion, 6 months, and  $1\ \text{year}$
- Bar deviation assessed digitally by STL file superimposition at 6 months and 1 year

## **Study Setting:**

Prosthodontics Department, Faculty of Dentistry, Tanta University, and CAD/CAM

# laboratory

## Ethical Consideration:

Informed consent will be obtained from all participants according to the guidelines of the Research Ethics Committee, Faculty of Dentistry, Tanta University

# Key References (Optional):

- 1. Resnik RR. Misch's Contemporary Implant Dentistry. 4th ed. Elsevier; 2020.
- 2. Abdullah A, Muhammed F, Zheng B, Liu Y. An Overview of CAD/CAM in Restorative Dentistry. Dent Mater J. 2018;7:1-10.
- 3. Elkady DM, El-Sherbini NN. Footprint of Different Bar Materials on Complete Overdenture Retention. ADJC. 2023;5:397-404.